CLINICAL TRIAL: NCT00646646
Title: The Effect of Sedation on Eye Movements
Acronym: Eye Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Michael Froelich, M.D, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: F050721005; K23RR021874-01A1 (NIH)
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Saccadic Eye Movements
Keywords: Sedation; Eye Movements
MeSH Terms: interventions — Propofol; Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- propofol (Active Comparator): active drug
  Interventions: Drug: propofol
- dexmedetomidine (Active Comparator): sedative
  Interventions: Drug: dexmedetomidine
- midazolam (Active Comparator): Sedative
  Interventions: Drug: Midazolam
- placebo (Placebo Comparator): placebo control
  Interventions: Drug: saline placebo

INTERVENTIONS:
Drug: propofol — sedative
  Arms: propofol
Drug: dexmedetomidine — Sedative
  Arms: dexmedetomidine
Drug: Midazolam — sedative
  Arms: midazolam
Drug: saline placebo — saline placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether sedation affects saccadic eye movements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, human volunteers, age 19-65.
* American Society of Anesthesiology (ASA) class I-II for inclusion criteria

Exclusion Criteria:

* Pregnancy
* Respiratory disease (severe asthma, emphysema)
* Cardiac disease (coronary artery disease, congestive heart failure)
* Symptomatic reflux disease
* Advanced rheumatic disease involving cervical spine
* Propofol or egg allergy
* Neurological disease (stroke, intracranial processes)
* Severe anemia

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- General Clinical Research Center, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was held at the Clinical Research Unit in Jefferson Towers. There were 65 participants recruited between March 28, 2008 and September 24, 2008. All participants signed a written informed consent and was verified to all the information pertaining to their participation in the study.
Pre-assignment Details: A physical examination of each participant was used to assess their success in the study. Participants were excluded if they did not meat the BMI weight requirement and/or wanted to be excluded from the study.
Groups:
- Dexmedetomidine: Sedative Drug 1
- Midazolam: Sedative Drug 2
- Propofol: Sedative Drug 3
Period: Overall Study
Arm/Group | Dexmedetomidine | Midazolam | Placebo | Propofol
Started | 15 | 15 | 15 | 20
Completed | 15 | 15 | 15 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dexmedetomidine: sedative
  dexmedetomidine : Sedative
- Midazolam: Sedative
  Midazolam : sedative
- Placebo: placebo control
  saline placebo : saline placebo
- Propofol: active drug
  propofol : sedative
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Midazolam | Placebo | Propofol | Total
Number analyzed (Participants) | 15 | 15 | 15 | 20 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 20 | 65
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (9.22109) | 32 (6.94879) | 34.93333 (11.09998) | 34.93333 (12.49838) | 33.16666 (2.09797)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 10 | 9 | 35
  Male | 6 | 8 | 5 | 11 | 30
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 20 | 65

OUTCOME MEASURES:

1. Primary Outcome: Dynamic Eye Movement Measures
Description: Change in Eye Movements Parameters
Time Frame: baseline to Sedation State (approx. 1 hr)
Measure: Mean (95% Confidence Interval); unit: (degrees/second)
Groups:
- Placebo: placebo
Arm/Group | Dexmedetomidine | Midazolam | Propofol | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 20
(degrees/second) | -25 [-35 to -14] | -115 [-126 to -103] | -90 [-101 to -79] | 10 [-77 to 57]

ADVERSE EVENTS:
Time Frame: The observation of adverse events will occur from the beginning of sedation monitoring up to discharge (1-4 hrs)
Arm/Group | Dexmedetomidine | Midazolam | Placebo | Propofol
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/20
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes